CLINICAL TRIAL: NCT05969041
Title: MYE Symphony: A Phase 1, Open-Label, First-in-Human, Dose Escalation Study to Investigate the Safety, Pharmacokinetics, Pharmacodynamics and Preliminary Efficacy of MT-302 in Adults With Advanced or Metastatic Epithelial Tumors
Brief Title: Study of MT-302 in Adults With Advanced or Metastatic Epithelial Tumors
Acronym: MYE Symphony
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Myeloid Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MTX-TROP2-302
Record Dates: First submitted 2023-07-06; First posted 2023-08-01 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Epithelial Tumors, Malignant
Keywords: Urothelial cancer; Cervical cancer; Ovarian epithelial; Triple-negative breast cancer; HR+/HER2- breast cancer; Pancreatic ductal adenocarcinoma; Gastric adenocarcinoma; Esophageal carcinoma; Non-small cell lung cancer; Colorectal cancer; TROP-2 expressing tumors; MT-302; Anti-TROP-2 chimeric antigen receptor; Myeloid cells; Monocytes; Chimeric Antigen Receptor (CAR); mRNA; Lipid nanoparticle (LNP)
MeSH Terms: conditions — Carcinoma; Uterine Cervical Neoplasms; Triple Negative Breast Neoplasms; Esophageal Neoplasms; Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A (MT-302) (Experimental): Participants will receive MT-302 through intravenous infusion.
  Interventions: Drug: MT-302 (A)

INTERVENTIONS:
Drug: MT-302 (A) — MT-302 is an investigational drug

SUMMARY:
MYE Symphony is a multicenter, open-label, Phase 1 first-in-human study to assess the safety, tolerability, and define the RP2D of MT-302 in participants with advanced epithelial cancer.

DETAILED DESCRIPTION:
The study has 4 Cohorts. Each Cohort has 4 Cycles. For Cohorts 1-3, the dosing regimen will be every 14 days for 3 doses, followed by administration once every 28 days for three doses. For Cohort 4, the dosing regimen will be modified. Participants will receive one dose of MT-302 every week for 3 doses, followed by administration once every 28 days for three additional doses.

A Safety Review Committee (SRC) will provide oversight for this study. The primary responsibility of the SRC is to safeguard study participants by reviewing and assessing the clinical safety data being collected during the conduct of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Adults age ≥ 18 inclusive at the time the Informed Consent Form (ICF) is signed.
2. Histologically proven, metastatic or advanced epithelial cancer including the following cancer types:

   1. Urothelial
   2. Cervical
   3. Ovarian epithelial
   4. Triple-negative breast
   5. HR+/HER2- breast
   6. Pancreatic ductal adenocarcinoma
   7. Gastric adenocarcinoma
   8. Esophageal carcinoma
   9. Non-small cell lung
   10. Colorectal
3. Progressive disease at baseline, refractory or relapsed to standard of care or who have declined standard therapy.
4. Measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) criteria v 1.1.
5. Eastern Cooperative Oncology Group (ECOG) performance status grade of 0 or 1.
6. Life expectancy of > 12 weeks.
7. Echocardiogram (ECHO) or multiple gated acquisition scan showing an ejection fraction greater than or equal to 50%.
8. Electrocardiogram (ECG) showing no clinically significant abnormality at Screening or showing an average QTc interval < 450 msec in males and < 470 msec in females (< 480 msec for participants with bundle branch block). Either Fridericia's or Bazett's formula may be used to correct the QT interval.
9. Oxygen saturation of greater than or equal to 90% on room air measured by pulse oximetry.
10. Adequate organ function as defined by laboratory values at Screening.
11. Willing and able to provide written informed consent.
12. Willing to perform and comply with all study procedures including undergoing study-related biopsies and attending clinic visits as scheduled.
13. Men must abstain from sperm donation during study treatment or for 4 months following last dose of study treatment.
14. Men and WOCBP must be willing to practice a highly effective method of contraception.

Exclusion Criteria:

1. Known active CNS metastasis and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, (ie, without evidence of progression for at least 4 weeks by repeat imaging), clinically stable, and without requirement of steroid treatment for at least 14 days prior to the first dose of study intervention.
2. Pregnant or nursing women.
3. Must be > 28 days beyond major surgery, including hepatectomy or joint replacement.
4. Prior allogeneic bone marrow transplantation or solid organ transplant.
5. Spinal cord compression not definitively treated with surgery and/or radiation.
6. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures.
7. Any acute illness including fever (> 100.4° F or > 38° C) within 7 days prior to Day 1
8. Active systemic bacterial, fungal, or viral infection within 7 days prior to Day 1. Participant cannot have tested positive for COVID-19 within 7 days prior to Day 1.
9. Active infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV), hepatitis C virus (HCV).
10. Other primary malignancies, except:

    1. Adequately treated basal cell or squamous cell carcinoma
    2. In situ carcinoma of the cervix or bladder, treated curatively and without evidence of recurrence for at least 2 years prior to the study, or
    3. A primary malignancy which has been completely resected and in complete remission for at least 2 years
11. History of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
12. Prior grade > 3 immune-related AEs such as pneumonitis, colitis, hepatitis, nephritis; prior dermatitis and endocrinopathies are allowed provided corticosteroids are no longer required and endocrine-replacement therapy is stable and discontinued from prior therapy.
13. Active autoimmune disease not related to prior therapy for primary malignancy that has required systemic therapy in the last 1 year.
14. History of symptomatic congestive heart failure (New York Heart Association classes II-IV) or serious active arrhythmias or other clinically significant cardiac disease within 12 months of enrollment.
15. Toxicity from previous anti-cancer therapy defined as toxicities (other than alopecia, or laboratory values listed above) not yet resolved to NCI CTCAE v5.0 Grade ≤ 1 or baseline. Participants with chronic Grade 2 toxicities (eg, peripheral neuropathy, laboratory values) may be eligible per the discretion of the Investigator and Medical Monitor.
16. Has received:

    1. Radiotherapy within 2 weeks of first administration of MT-302
    2. Cytotoxic chemotherapy for treatment of the primary malignancy within 28 days or 5 half-lives, whichever is shorter, of administration of MT-302
    3. Immune therapy for primary malignancy (eg, monoclonal antibody therapy, checkpoint inhibitors) within 28 days or 5 half-lives, whichever is shorter of first administration of MT-302
    4. Targeted therapies for primary malignancy within 28 days or 5 half-lives, whichever is shorter, of first administration of MT-302
    5. Anti-cancer vaccine within 12 weeks of first administration of MT-302
    6. COVID-19 mRNA vaccine within 6 weeks of first administration of MT-302
17. Has received a live vaccine ≤ 6 weeks prior to first administration of MT-302
18. Has received packed red blood cells or platelet transfusion within 2 weeks prior to first administration of MT-302
19. History of an allergic reaction to any of the excipients
20. Enrollment in another interventional clinical trial within 28 days or 5 half-lives of the drug, whichever is shorter, of first administration of MT-302
21. Any other condition that, in the opinion of the Investigator, would make the participant unsuitable for the study or unable to comply with the study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-08-02 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of MT-302 through incidence of Adverse Events | Up to Week 20
  Adverse Events will be graded according to the NCI-CTCAE, version 5.0
To establish the maximum tolerated dose (MTD) | Up to Week 20
  based on dose limiting toxicities (DLTs) and the recommended Phase 2 dose (RP2D)

SECONDARY OUTCOMES:
To further characterize the safety of MT-302 through incidence of Adverse Events | Up to Week 20
  Adverse Events will be graded according to the NCI-CTCAE, version 5.0
To assess the pharmacokinetics (PK) of MT-302 | Up to Week 20
  PK parameter: Plasma concentrations
To assess the pharmacokinetics (PK) of MT-302 | Up to Week 20
  PK parameter: Area under curve (AUC0-last, AUC 0-∞)
To assess the pharmacokinetics (PK) of MT-302 | Up to Week 20
  PK parameter: Time of maximum observed plasma concentration (tmax)
To assess the pharmacokinetics (PK) of MT-302 | Up to Week 20
  PK parameter: Apparent terminal Half-life (t1/2)
To assess the pharmacokinetics (PK) of MT-302 | Up to Week 20
  PK parameter: Plasma Clearance (CL)
To assess the pharmacokinetics (PK) of MT-302 | Up to Week 20
  PK parameter: Volume of Distribution (Vd)
To assess the pharmacokinetics (PK) of MT-302 | Up to Week 20
  PK parameter:Mean residence time (MRT)
To assess the pharmacokinetics (PK) of MT-302 | Up to Week 20
  PK parameter: terminal rate constant ( λz)
Determine rate of ICANS | Up to Week 20
  For grading of potential immune effector cell-associated neurotoxicity syndrome (ICANS), use of the 10-point immune effector cell-associated encephalopathy (ICE) screening tool
Determine rate of Grade 3-5 CRS | Up to Week 20
  ASCO CRS Grading

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Maurer, MD, Study Director — Myeloid Therapeutics
Locations (6):
- Australia (6):
  - St Vincent's Public Hospital Sydney, Darlinghurst, New South Wales
  - Scientia Clinical Research Ltd, Randwick, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Souther Oncology Clinical Research Unit (SOCRU), Bedford Park, South Australia
  - Cabrini Health, Malvern, Victoria
  - Linear Clinical Research Ltd, Nedlands, Western Australia